CLINICAL TRIAL: NCT01134458
Title: Personalized Cardiovascular Risk Information to Initiate and Maintain Health Behavior Changes
Acronym: FIMDM_CVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00024341; FIMDM Research Grant 0170-1 (Other Grant/Funding Number: Foundation for Informed Medical Decision Making, Inc)
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Cardiovascular Disease; Peripheral Artery Disease; Ischemic Stroke; Diabetes
Keywords: cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Peripheral Arterial Disease; Ischemic Stroke; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Receive primary care and management of CVD according to the discretion of their primary care provider. They will also receive generic educational information concerning CVD at baseline and at study end (at their request). We will collect outcomes at baseline and 3-months.
- Web-based Intervention (Experimental): Given current risk assessment for CVD based on Health Dialog Cardiac Risk Calculator, recommendations for behavior change, and Health Dialog's Living with Coronary Heart Disease. Can change initial patient risk information provided by the Risk Calculator during the initial visit, noting what they are will work on during the study. Sent monthly email reminders to log onto the system to choose that months' behavioral modules. Given a choice of at least 2 health behavior modules per month (smoking cessation, exercise, diet, and weight) to improve their CVD risk. Information on risk, CVD knowledge, medication management and side effects will be provided to all participants. It will also provide tailored information to help the individual initiate and maintain these behaviors.
  Interventions: Behavioral: Web-Based Intervention

INTERVENTIONS:
Behavioral: Web-Based Intervention — 1. Health Dialog Cardiac Risk Calculator
  2. Health Dialog's Living with Coronary Heart Disease
  3. Tailored intervention including health behavior modules such as smoking cessation, exercise, diet, and weight
  Other Names: Health Dialog Cardiac Risk Calculator
  Arms: Web-based Intervention

SUMMARY:
The investigators propose an evaluation that will assess three important components of risk communication:

1. provide patients with personalized risk communication using the risk calculator developed by FIMDM and health information taken from the Living with Coronary Artery Disease program
2. provide personalized tailored patient feedback to help initiate and maintain specific cardiovascular CVD-related behaviors(e.g., medication adherence, exercise, diet, smoking cessation) to reduce their risks.
3. evaluate how this feedback can be incorporated into clinical care by examining 3 month patient outcome and provider responses to the risk information.

DETAILED DESCRIPTION:
Patients at high risk for CVD events frequently underestimate their risk. Programs to improve CVD outcomes have largely focused on single risk factors and do not contextualize the information with a patient's global risk. An easy, accessible strategy to address global CVD risk based on personalized risk communication feedback with assistance with initiating and maintaining health behaviors has several advantages, but has not formally been tested. A patient's perceived risk of stroke or heart attack is an important factor in understanding motivation for risk reducing behaviors. Lower perceived risk has been associated with poorer adherence to recommended health behaviors. Additionally, a person's beliefs about his or her risk for a disease increased the likelihood of a more informed and activated patient, and figures prominently in models of health behavior (e.g., Health Belief Model). People tend to underestimate their own risk; Therefore providing accurate risk communication has the potential to activate patients to initiate and maintain behavior changes.

ELIGIBILITY:
Inclusion Criteria:

* cardiovascular disease (CVD)
* CVD risk equivalent (peripheral arterial disease, history of ischemic stroke, or diabetes)

Exclusion Criteria:

* metastatic cancer,
* dementia,
* active psychosis
* end-stage renal disease
* no access to computer with Internet

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Disease (CVD) Risk Knowledge Assessment | Baseline and 3 month @ study end
  Trained personnel will obtain the patients' outcome values (i.e., weight, height, BP) at baseline and subsequent 3-month outcome using a digital sphygmomanometer and digital scale according to a standard protocol. The baseline interview includes demographics and an assessment of patients' health behavior, perceived risk, and interactions with their provider. At 3-month follow-up visit, patients will also undergo an in-person interview to determine changes in weight, smoking status, medication adherence, decisional conflict, knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Hayden Bosworth, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States